CLINICAL TRIAL: NCT07182201
Title: Effect of Foot Core Control Training on Dorsiflexion Function and Gait Biomechanical Characteristics of Patients With Chronic Plantar Fasciitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20250140
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Plantar Fasciitis; Functional Hallux Limitus
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot core control training combined + regular CPF training (Experimental)
  Interventions: Behavioral: Foot core control training; Behavioral: CPF Conventional training
- regular CPF training (Active Comparator)
  Interventions: Behavioral: CPF Conventional training

INTERVENTIONS:
Behavioral: Foot core control training — (1) Toe Yoga : When MTPJ1 actively dorsiflexes, the other four toes remain in contact with the ground. The subject lifts the big toe while the remaining four toes stay on the ground; conversely, when the big toe contacts the ground, the other four toes lift upward, alternating this pattern. (2)Doming: While keeping MTPJ1 in contact with the ground, elevate the foot arch. This exercise strengthens intrinsic foot muscle strength, helping stabilize the arch and first metatarsal. The subject tightens the toes, bringing the forefoot toward the heel to form and enhance the arch. Maintain all toes firmly planted on the ground, ensuring no ankle inversion, no forced flexion or extension of toes, and hold at maximum position. Perform training seated to avoid compensatory movements by external muscles during exercise. (3) Toe Abduction Exercises（4）Dynamic Exercise Progression
  Arms: Foot core control training combined + regular CPF training
Behavioral: CPF Conventional training — The key points of the exercise are as follows: (1) Fascia ball release of plantar fascia (2) Plantar fascia stretching (3) Gastrocnemius muscle stretching (4) Toe grab towel

SUMMARY:
The pain and abnormal gait postures observed in CPF patients may be associated with impaired foot function. However, few studies have examined the dorsiflexion function of the big toe in CPF patients, and the effectiveness of foot core control training in alleviating pain and improving gait remains unclear. Restricted movement of the metatarsophalangeal joint (MTPJ1) may severely compromise foot function, leading to gait pattern alterations and subsequent instability. To address this, our study aims to improve symptoms, functional outcomes, and gait through foot core control training interventions. We recorded kinematic parameters and biomechanical data during the foot's plantar phase at toe-off before and after functional training for CPF patients. Comparative analysis between intervention groups revealed whether foot core control training can effectively enhance big toe dorsiflexion function and gait biomechanics in CPF patients. This research clarifies the therapeutic efficacy of foot core control training for CPF patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Ultrasound findings indicating plantar fascia thickness>4 mm or 20% thickening compared to the contralateral side; (2) Age 25-45 years; (3) Ankle dorsiflexion range <65° in weight-bearing standing position; (4) Persistent heel pain lasting ≥3 months but ≤1 year; (5) No prior treatment within 1 month prior to hospital admission; (6) Subjects without prior CPF surgical intervention.

Exclusion Criteria:

* (1) Concurrent presence of severe malignant diseases; (2) Abnormal conditions such as skin ulcers or infections on the sole; (3) Concurrent neurological or immunological disorders; (4) Concurrent heel deformity or fracture; (5) Secondary CPF caused by rheumatoid arthritis, ankylosing spondylitis, or other conditions; (6) Concurrent cognitive impairment, mental abnormalities, or difficulty completing relevant assessment scales.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vicon 3D gait test | 30 minutes
  subjects wore athletic shorts, fully exposing the waist and the area below the mid-thigh. After reflective markers were attached, subjects familiarized themselves with the movement collection requirements and procedures according to the testing protocol. They stood in the center of the testing room with their feet shoulder-width apart and upper limbs resting naturally at their sides, maintaining the subtalar joint in a neutral position. A static test was conducted to collect reference data for defining the coordinate systems of the bone segments. Subsequently, participants performed walking, jogging, side-cutting, jumping, and single-leg balance tasks at a self-selected comfortable pace. Sufficient rest was provided between trials to prevent fatigue. Five valid trials were collected for each movement, and the average of three trials was used for analysis.
Evaluation of dorsiflexion function of big toe | 30 minutes
  Goniometric measurement: The subject removes footwear and stands weight-bearing on a yoga mat, actively dorsiflexing the big toe. The tester measures the dorsiflexion angle of the big toe using a goniometer. The goniometer's axis is aligned with the big toe's MTPJ1, with the fixed arm parallel to the first metatarsal and the movable arm parallel to the first proximal phalanx. The movable arm is adjusted according to the subject's dorsiflexion angle, with measurements recorded. Three trials are performed and averaged.
  Vicon measurement: The subject's MTPJ1 angle during walking is recorded using Vicon technology.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 5minutes
ankle and hindfoot function scale (AOFAS) | 5 minutes

IPD SHARING:
Plan to Share IPD: No